CLINICAL TRIAL: NCT04647526
Title: A Phase 3, Open-Label, Randomized Study Evaluating Metastatic Castrate Resistant Prostate Cancer Treatment Using PSMA [Lu-177]-PNT2002 Therapy After Second-line Hormonal Treatment (SPLASH)
Brief Title: Study Evaluating mCRPC Treatment Using PSMA [Lu-177]-PNT2002 Therapy After Second-line Hormonal Treatment
Acronym: SPLASH
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: POINT Biopharma, a wholly owned subsidiary of Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27232; J5T-OX-JXCA (Other: Eli Lilly and Company); PBP-301 (Other: POINT Biopharma Global Inc); 2021-002641-15 (EudraCT Number); 2024-515604-39-00 (EU CTIS Number)
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Results first posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer
Keywords: PSMA; mCRPC; Prostate cancer; 177Lu-PSMA; radioligand therapy; PSMA-I&T; SPLASH
MeSH Terms: conditions — Prostatic Neoplasms | interventions — abiraterone; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Lead-in Dosimetry Phase: [Lu-177]-PNT2002 (Experimental): Participants received 6.8 gigabecquerels (GBq) (±10%) of [Lu-177]-PNT2002 by intravenous infusion every 8 weeks for 4 cycles.
  Interventions: Drug: [Lu-177]-PNT2002
- Randomization Phase: [Lu-177]-PNT2002 (Arm A) (Experimental): Participants received 6.8 GBq (±10%) of [Lu-177]-PNT2002 by intravenous infusion every 8 weeks for 4 cycles.
  Interventions: Drug: [Lu-177]-PNT2002
- Randomization Phase: Abiraterone or Enzalutamide (Arm B) (Active Comparator): Participants received either of below treatments until radiographic progression.
  * Enzalutamide 160 milligram (mg) orally once daily (or)
  * Abiraterone 1000 mg orally once daily coadministered with prednisone 5 mg orally twice daily or dexamethasone 0.5 mg orally once daily.
  Participants who experienced radiographic progression per Blinded Independent Central Review (BICR) (or after final overall survival (OS), per local investigator-assessment), had not started an intervening treatment, and had no uncontrolled adverse events (AEs) were eligible to consent to cross over to receive 6.8 GBq (±10%) of [Lu-177]-PNT2002 intravenous infusion every 8 weeks for 4 cycles.
  Interventions: Drug: [Lu-177]-PNT2002; Drug: Abiraterone; Drug: Enzalutamide
- Pharmacokinetic (PK) Extension Phase: [Lu-177]-PNT2002 (Experimental): Participants received 6.8 GBq (±10%) of [Lu-177]-PNT2002 by intravenous infusion every 8 weeks for 4 cycles.
  Interventions: Drug: [Lu-177]-PNT2002

INTERVENTIONS:
Drug: [Lu-177]-PNT2002 — Participants randomized to Arm A will receive 6.8 GBq (±10%) of [Lu-177]-PNT2002 every 8 weeks for 4 cycles
  Other Names: [Lu-177]-PSMA-I&T; LY4187525
Drug: Abiraterone — Abiraterone (1000 mg orally once daily with: 5 mg twice daily prednisone or 0.5 mg once daily dexamethasone)
  Arms: Randomization Phase: Abiraterone or Enzalutamide (Arm B)
Drug: Enzalutamide — Enzalutamide (160 mg orally once daily)
  Arms: Randomization Phase: Abiraterone or Enzalutamide (Arm B)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of [Lu-177]-PNT2002 in patients with metastatic castration-resistant prostate cancer who have progressed following treatment with androgen receptor axis-targeted therapy (ARAT).

DETAILED DESCRIPTION:
The primary objective of the study is to determine the efficacy of [Lu-177]-PNT2002 ([Lu-177]-PSMA-I&T) versus abiraterone or enzalutamide in delaying radiographic progression in patients with mCRPC.

The study consists of 3 phases: Dosimetry, Randomized Treatment, and Long term Follow up.

The study will commence with a 25-patient safety and dosimetry lead-in (Part 1) and proceed to a randomization treatment phase in approximately 390 patients (Part 2). Patients in Part 2 will be randomized in a 2:1 ratio to receive either [Lu-177]-PNT2002 (Arm A), or enzalutamide or abiraterone (Arm B). Patients in Arm B who experience radiographic progression per central review and meet protocol defined eligibility, may crossover to receive [Lu-177]-PNT2002. After final overall survival (OS) analysis, all patients will continue to be followed through Continued Access, including long-term follow-up (LTFU) for at least 5 years from the first therapeutic dose, death, or loss to follow up (Part 3).

Only patients that meet PSMA PET avidity criteria per central review will be eligible for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male aged 18 years or older.
2. Histological, pathological, and/or cytological confirmation of adenocarcinoma of the prostate.
3. Ineligible or averse to chemotherapeutic treatment options.
4. Patients must have progressive mCRPC at the time of consent based on at least 1 of the following criteria:

   1. Serum/plasma PSA progression defined as increase in PSA greater than 25% and >2 ng/mL above nadir, confirmed by progression at 2 time points at least 3 weeks apart.
   2. Soft-tissue progression defined as an increase ≥20% in the sum of the diameter (SOD) (short axis for nodal lesions and long axis for non-nodal lesions) of all target lesions based on the smallest SOD since treatment started or the appearance of one or a new lesion.
   3. Progression of bone disease defined as the appearance of two or more new lesions by bone scan.
5. Progression on previous treatment with one ARAT (abiraterone or enzalutamide or darolutamide or apalutamide) in either the CSPC or CRPC setting.
6. PSMA-PET scan (i.e., 68Ga-PSMA-11 or 18F-DCFPyL) positive as determined by the sponsor's central reader.
7. Castrate circulating testosterone levels (<1.7 nmol/L or <50 ng/dL).
8. Adequate organ function, independent of transfusion:

   1. Bone marrow reserve:

      * i. White blood cell (WBC) count ≥2.5 × 10^9/L OR absolute neutrophil count (ANC) ≥1.5 × 10^9/L.
      * ii. Platelets ≥100 × 10^9/L.
      * iii. Hemoglobin ≥8 mmol/L.
   2. Liver function:

      * i. Total bilirubin ≤1.5 × institutional upper limit of normal (ULN). For patients with known Gilbert's syndrome, ≤3 × ULN is permitted.
      * ii. ALT or AST ≤3.0× ULN.
   3. Renal function:

      * i. Serum/plasma creatinine ≤1.5 × ULN or creatinine clearance ≥50 mL/min based on Cockcroft-Gault formula (for patients in France, serum/plasma creatinine ≤1.5 × ULN or CrCl ≥60 mL/min based on Cockcroft-Gault formula).
   4. Albumin ≥30 g/L.
9. Human immunodeficiency virus-infected patients who are healthy and have a low risk of acquired immunodeficiency syndrome-related outcomes are included in this trial.
10. For patients who have partners who are pregnant or of childbearing potential: a condom is required along with a highly effective contraceptive method during the study and for 6 months after last study drug administration. Such methods deemed highly effective include a) combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation, b) progestogen-only hormonal contraception associated with inhibition of ovulation, c) intrauterine device (IUD), d) intrauterine hormone-releasing system (IUS), e) bilateral tubal occlusion, f) vasectomy, g) true sexual abstinence: when this is in line with the preferred and usual lifestyle of the subject [periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of exposure to IMP, and withdrawal are not acceptable methods of abstinence].
11. Willing to initiate ARAT therapy (either enzalutamide or abiraterone), pre-specified by investigator, if randomized to Treatment Arm B.
12. ECOG performance status 0 to 1.
13. Willing and able to comply with all study requirements and treatments (including 177Lu PNT2002) as well as the timing and nature of required assessments.
14. Signed informed consent.

Exclusion Criteria:

Patients are excluded from the study if any of the following criteria apply:

1. If noted in pathology report, prostate cancer with known significant (>10% present in cells) sarcomatoid or spindle cell or neuroendocrine components. Any small cell component in the cancer should result in exclusion.
2. Prior treatment for prostate cancer ≤28 days prior to randomization, with the exclusion of first-line local external beam, ARAT, luteinizing hormone-releasing hormone (LHRH) therapy, or non-radioactive bone-targeted agents.
3. Any prior cytotoxic chemotherapy for CRPC (e.g., cabazitaxel or docetaxel); chemotherapy for hormone-sensitive prostate cancer (HSPC) is allowed if the last dose was administered >1 year prior to consent.
4. Prior treatment with systemic radionuclides (e.g. radium-223, rhenium-186, strontium 89).
5. Prior immuno-therapy, except for sipuleucel-T.
6. Prior PSMA-targeted radioligand therapy, e.g., Lu-177-PSMA-617, I 131-1095.
7. Prior poly ADP ribose polymerase (PARP) inhibitor for prostate cancer.
8. Patients who progressed on 2 or more lines of ARATs.
9. Patients receiving bone-targeted therapy (e.g. denosumab, zoledronic acid) not on stable doses for at least 4 weeks prior to randomization.
10. Administration of an investigational agent ≤60 days or 5 half-lives, whichever is shorter, prior to randomization.
11. Major surgery ≤30 days prior to randomization.
12. Estimated life expectancy <6 months as assessed by the principal investigator.
13. Presence of liver metastases >1 cm on abdominal imaging.
14. A superscan on bone scan defined as a bone scan that demonstrates markedly increased skeletal radioisotope uptake relative to soft tissues in association with absent or faint genitourinary tract activity.
15. Dose escalation or initiation of opioids for cancer-related pain ≤30 days prior to consent up to and including randomization.
16. Known presence of central nervous system metastases.
17. Contraindications to the use of planned ARAT therapy, [Ga-68]-PSMA-11, [F-18]-DCFPyL or [Lu-177]-PNT2002 therapy, including but not limited to the following:

    * Hypersensitivity to [Ga-68]-PSMA-11, [F-18]-DCFPyL or [Lu-177]-PNT2002 excipients (Diethylenetriaminepentaacetic acid (DTPA), Sodium ascorbate, Lascorbic acid, Sodium gentisate, HCl, Sodium hydroxide).
    * Recent myocardial infarction or arterial thrombotic events (in the past 6 months) or unstable angina (in the past 3 months), bradycardia or left ventricular ejection fraction measurement of < 50%.
    * History of seizures in patients planned to receive enzalutamide.
18. Active malignancy other than low-grade non-muscle-invasive bladder cancer and non-melanoma skin cancer.
19. Concurrent illness that may jeopardize the patient's ability to undergo study procedures.
20. Serious psychological, familial, sociological, or geographical condition that might hamper compliance with the study protocol and follow-up schedule. Patients that travel need to be capable of repeated visits even if they are on the control arm.
21. Symptomatic cord compression, or clinical or radiologic findings indicative of impending cord compression.
22. Concurrent serious (as determined by the investigator) medical conditions, including, but not limited to, New York Heart Association class III or IV congestive heart failure (see 12.1 Appendix 1), unstable ischemia, uncontrolled symptomatic arrhythmia, history of congenital prolonged QT syndrome, uncontrolled infection, known active hepatitis B or C, or other significant co-morbid conditions that in the opinion of the investigator would impair study participation or cooperation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2028-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Jensen, Study Director — Eli Lilly and Company
Locations (54):
- United States (33):
  - Arizona Institute of Urology (AIU) - Tucson, Tucson, Arizona
  - Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - University of California Los Angeles, Nuclear Medicine Clinic, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - UC Irvine Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute, Palo Alto, California
  - University of Colorado Hospital, Aurora, Colorado
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Tulane University Medical Center, New Orleans, Louisiana
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Chesapeake Urology Associates (CUA) P.A., Towson, Maryland
  - University of Michigan Hospitals, Ann Arbor, Michigan
  - Karmanos Cancer Center, Detroit, Michigan
  - VA St. Louis Health Care System, St Louis, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Urology Cancer Center, PC, Omaha, Nebraska
  - Astera Cancer Care, East Brunswick, New Jersey
  - New Mexico Oncology Hematology Consultants Ltd., New Mexico Cancer Center, Albuquerque, New Mexico
  - New York Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - Tri-State Urologic Services, Cincinnati, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Dallas VA Medical Center, Nuclear Medicine Service, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Excel Diagnostics & Nuclear Oncology Center, Houston, Texas
  - Swedish Cancer Institute Research, Seattle, Washington
- Canada (8):
  - BC Cancer - Vancouver, Vancouver, British Columbia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - London Health Sciences Center - Victoria Hospital, London, Ontario
  - Sunnybrook Research Institute, Odette Cancer Center, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - CHUM - University Hospital of Montreal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHU of Quebec - Laval University, Québec, Quebec
- France (6):
  - Center Jean Perrin, Department of Medical Oncology, Clermont-Ferrand
  - Claude Huriez Hospital, Lille
  - Leon Berard Center, Lyon
  - La Timone Hospital, Nuclear Medicine Department, Marseille
  - Montpellier Cancer Institute, Department of Nuclear Medicine, Montpellier
  - Tenon Hospital, Department of Medical Oncology, Paris
- Netherlands (3):
  - St. Antonius Hospital, Nieuwegein
  - Radboud University Medical Center (Radboudumc), Nijmegen
  - Erasmus University Medical Center Rotterdam, Rotterdam
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Norrlands University Hospital, Department of Radiation Sciences, Oncology, Umeå
- United Kingdom (2):
  - Charing Cross Hospital, Department of Medical Oncology, London
  - Royal Marsden NHS Foundation Trust - Institute of Cancer Research, Sutton

REFERENCES:
- [Background] Baum RP, Kulkarni HR, Schuchardt C, Singh A, Wirtz M, Wiessalla S, Schottelius M, Mueller D, Klette I, Wester HJ. 177Lu-Labeled Prostate-Specific Membrane Antigen Radioligand Therapy of Metastatic Castration-Resistant Prostate Cancer: Safety and Efficacy. J Nucl Med. 2016 Jul;57(7):1006-13. doi: 10.2967/jnumed.115.168443. Epub 2016 Jan 21. PMID 26795286
- [Derived] Hansen AR, Probst S, Beauregard JM, Viglianti BL, Michalski JM, Tagawa ST, Sartor O, Tutrone RF, Oz OK, Courtney KD, Delpassand ES, Nordquist LT, Osman MM, Chi KN, Sparks R, George N, Hawley SM, Wu W, Jensen JD, Fleshner NE. Initial clinical experience with [177Lu]Lu-PNT2002 radioligand therapy in metastatic castration-resistant prostate cancer: dosimetry, safety, and efficacy from the lead-in cohort of the SPLASH trial. Front Oncol. 2025 Jan 7;14:1483953. doi: 10.3389/fonc.2024.1483953. eCollection 2024. PMID 39839782
- [Derived] American College of Nuclear Medicine (ACNM) 2022 ACNM Annual Meeting AbstractsJanuary 27-29, 2022 Virtual Meeting. Clin Nucl Med. 2023 Feb 3:e246-e277. doi: 10.1097/RLU.0000000000004535. Online ahead of print. No abstract available. PMID 36735603
- See also: 1400P - Efficacy and safety of 177Lu-PNT2002 prostate-specific membrane antigen (PSMA) therapy in metastatic castration resistant prostate cancer (mCRPC): Initial results from SPLASH — https://cslide.ctimeetingtech.com/esmo2022/attendee/confcal_2/presentation/list?q=1400P
- See also: ESMO 2024: Efficacy of 177Lu-PNT2002 in PSMA-Positive mCRPC Following Progression on an Androgen-Receptor Pathway Inhibitor (SPLASH) — https://www.urotoday.com/conference-highlights/esmo-2024/esmo-2024-prostate-cancer/154850-esmo-2024-efficacy-of-177lu-pnt2002-in-psma-positive-mcrpc-following-progression-on-an-androgen-receptor-pathway-inhibitor-splash.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study includes:
  * Lead-in dosimetry phase to evaluate the dosimetry of [Lu-177]-PNT2002 across standard organs such as the kidneys, salivary and lacrimal glands.
  * Randomization phase to compare the efficacy of [Lu-177]-PNT2002 versus enzalutamide or abiraterone (control arm).
  Additionally, there is a pharmacokinetic (PK) extension phase, in which participants were enrolled at selected sites in the United States and Canada for PK assessments of [Lu-177]-PNT2002.
Pre-assignment Details: (continued.,) Participants were unique to each phase of the study, those participated in one phase did not transition to any other phase. All participants will be followed in the long-term follow-up phase for at least five years from the date of their first therapeutic dose, or until death or loss to follow-up, whichever occurs first.
Groups:
- PK Extension Phase: [Lu-177]-PNT2002: Participants received 6.8 GBq (±10%) of [Lu-177]-PNT2002 by intravenous infusion every 8 weeks for 4 cycles.
Period: Overall Study
Arm/Group | Lead-in Dosimetry Phase: [Lu-177]-PNT2002 | Randomization Phase: [Lu-177]-PNT2002 (Arm A) | Randomization Phase: Abiraterone or Enzalutamide (Arm B) | PK Extension Phase: [Lu-177]-PNT2002
Started | 27 | 276 | 136 | 16
Intent-to-Treat Analysis (ITT) Set (All participants who were randomly assigned to Arm A or Arm B, regardless of the treatment they actually received.) | 0 (This milestone is not applicable for this arm.) | 276 | 136 (As per the prespecified statistical analysis plan, the efficacy analysis for Arm B was conducted as a whole, regardless of whether participants received Abiraterone or Enzalutamide, or crossed over to [Lu-177]-PNT2002.) | 0 (This milestone is not applicable for this arm.)
Participants on Arm B Treatment Who Crossed Over to [Lu-177]-PNT2002 | 0 (This milestone is not applicable for this arm.) | 0 (This milestone is not applicable for this arm.) | 77 | 0 (This milestone is not applicable for this arm.)
Safety Analysis Set (All participants who received at least one dose of the study drug.) | 27 | 269 | 130 (As per the prespecified statistical analysis plan, safety analysis for Arm B was conducted as a whole, regardless of whether participants received Abiraterone or Enzalutamide. Additionally, safety data for the crossover group were planned to be reported separately. * Participants who received at least one dose of Abiraterone or Enzalutamide = 130 * Participants who crossed over and received at least one dose of [Lu-177]-PNT2002 = 77) | 15
Completed (Participants who completed the 5-year follow-up are considered study completers.) | 0 | 0 | 0 | 0
Not Completed | 27 | 276 | 136 | 16
Not completed — Death | 13 | 76 | 32 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 15 | 8 | 1
Not completed — Incorrect enrollment | 0 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 1 | 0
Not completed — Ongoing | 9 | 183 | 93 | 15

BASELINE CHARACTERISTICS:
Population: All participants in the study.
Groups:
- Lead-in Dosimetry Phase: [Lu-177]-PNT2002; Randomization Phase: [Lu-177]-PNT2002 (Arm A); PK Extension Phase: [Lu-177]-PNT2002: Participants received 6.8 GBq (±10%) of [Lu-177]-PNT2002 by intravenous infusion every 8 weeks for 4 cycles.
- Randomization Phase: Abiraterone or Enzalutamide (Arm B): Participants received either of below treatments until radiographic progression.
  * Enzalutamide 160 mg orally once daily (or)
  * Abiraterone 1000 mg orally once daily coadministered with prednisone 5 mg orally twice daily or dexamethasone 0.5 mg orally once daily.
  Participants who experienced radiographic progression per BICR (or after final OS, per local investigator-assessment), had not started an intervening treatment, and had no uncontrolled AEs were eligible to consent to cross over to receive 6.8 GBq (±10%) of [Lu-177]-PNT2002 intravenous infusion every 8 weeks for 4 cycles.
- Total: Total of all reporting groups
Arm/Group | Lead-in Dosimetry Phase: [Lu-177]-PNT2002 | Randomization Phase: [Lu-177]-PNT2002 (Arm A) | Randomization Phase: Abiraterone or Enzalutamide (Arm B) | PK Extension Phase: [Lu-177]-PNT2002 | Total
Number analyzed (Participants) | 27 | 276 | 136 | 16 | 455
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 52 | 27 | 0 | 86
  >=65 years | 20 | 224 | 109 | 16 | 369
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 27 | 276 | 136 | 16 | 455
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 5 | 1 | 9
  Not Hispanic or Latino | 26 | 262 | 129 | 15 | 432
  Unknown or Not Reported | 0 | 12 | 2 | 0 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 11 | 2 | 0 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 32 | 8 | 1 | 45
  White | 23 | 215 | 112 | 15 | 365
  More than one race | 0 | 2 | 2 | 0 | 4
  Unknown or Not Reported | 0 | 16 | 12 | 0 | 28
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 12 | 78 | 42 | 1 | 133
  Netherlands | 0 | 11 | 6 | 0 | 17
  Sweden | 0 | 3 | 5 | 0 | 8
  United States | 15 | 149 | 65 | 15 | 244
  United Kingdom | 0 | 10 | 3 | 0 | 13
  France | 0 | 25 | 15 | 0 | 40

OUTCOME MEASURES:

1. Primary Outcome: Randomization Phase: Radiographic Progression-Free Survival (rPFS)
Description: * rPFS, as assessed by blinded independent central review (BICR), is the time from the randomization date to progression on soft tissue per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) or confirmed progression on bone lesions by Prostate Cancer Working Group 3 (PCWG3) criteria, or death from any cause.
  * The date of disease progression is the date of the scan for the first objectively documented progressive disease (PD) per RECIST v1.1 or PCWG3. PD is defined as a ≥20% increase in the sum of the diameters of target lesions (≥5 mm absolute), with reference being the smallest sum in the study, or unequivocal progression of non-target lesions, or appearance of new lesions.
  * Participants who do not progress, including those who started new anticancer therapy, withdrew from the study, or were lost to follow-up without disease progression, were censored at the last valid assessment for RECIST v1.1 or PCWG3.
Time Frame: From the randomization date to the first documented progressive disease or death from any cause (up to 23 months)
Population: All participants from the ITT analysis set. Number of participants censored in [Lu-177]-PNT2002 (Arm A)=114, Abiraterone or Enzalutamide (Arm B)=40. The "Overall Number of Participants Analyzed" reported is inclusive of the censored participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomization Phase: [Lu-177]-PNT2002 (Arm A) | Randomization Phase: Abiraterone or Enzalutamide (Arm B)
Number analyzed (Participants) | 276 | 136
months | 9.5 [7.4 to 10.0] | 6.0 [4.7 to 7.9]
Statistical Analysis 1: Comparison: Randomization Phase: [Lu-177]-PNT2002 (Arm A) vs Randomization Phase: Abiraterone or Enzalutamide (Arm B); Test type: Superiority; p = 0.0088, Log Rank; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.55 to 0.92]

2. Secondary Outcome: Randomization Phase: Percentage of Participants With Objective Response Rate (ORR)
Description: * ORR, as assessed by BICR, is the best confirmed overall tumor response of complete response (CR) or partial response (PR) as per RECIST v1.1 ( in the absence of confirmed progression on bone scan assessed by PCWG3).
  * CR is a disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 millimeters (mm).
  * PR is at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters), without progression of non-target lesions or appearance of new lesions.
Time Frame: Randomization until measured progressive disease (up to 23 months)
Population: All participants from the ITT analysis set who had measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Randomization Phase: [Lu-177]-PNT2002 (Arm A) | Randomization Phase: Abiraterone or Enzalutamide (Arm B)
Number analyzed (Participants) | 97 | 50
percentage of participants | 32.0 [22.9 to 42.2] | 8.0 [2.2 to 19.2]

3. Secondary Outcome: Randomization Phase: Duration of Response
Description: Duration of Response, as assessed by BICR, is the time from the date of first documented confirmed CR or PR as per RECIST v1.1 (in the absence of confirmed progression on bone scan assessed by PCWG3) to the date of first documented radiographic progression or death in the absence of progression. Participants who have attained CR or PR as the best overall response, did not have progressive disease, and did not die will be censored.
Time Frame: From the date of first CR or PR to disease progression or death (up to 16.3 months)
Population: All participants from the ITT analysis set who had achieved confirmed CR or PR responses (ORR). Number of participants censored in [Lu-177]-PNT2002 (Arm A)=18, Abiraterone or Enzalutamide (Arm B)=1. The "Overall Number of Participants Analyzed" reported is inclusive of the censored participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomization Phase: [Lu-177]-PNT2002 (Arm A) | Randomization Phase: Abiraterone or Enzalutamide (Arm B)
Number analyzed (Participants) | 31 | 4
months | 9.4 [7.6 to 15.0] | 8.3 [4.0 to NA] — There were not enough events to estimate the upper limit of the 95% confidence interval.

4. Secondary Outcome: Randomization Phase: Percentage of Participants With Prostate-Specific Antigen (PSA) Response Rate
Description: The PSA response rate, as per the PCWG3 criteria, is the percentage of participants achieving a ≥50% decrease in PSA from baseline to the lowest post-baseline PSA result, confirmed by a second PSA assessment conducted at least 3 weeks later.
Time Frame: From the randomization up to 23 months
Population: All participants from the ITT analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Randomization Phase: [Lu-177]-PNT2002 (Arm A) | Randomization Phase: Abiraterone or Enzalutamide (Arm B)
Number analyzed (Participants) | 276 | 136
percentage of participants | 30.1 [24.7 to 35.9] | 12.5 [7.5 to 19.3]

5. Secondary Outcome: Randomization Phase: Biochemical Progression-Free Survival (bPFS)
Description: bPFS is the time from the date of randomization to the date of the first PSA increase from baseline ≥25% and ≥2 nanograms per milliliter (ng/mL) above nadir confirmed by a second PSA measurement defining progression ≥3 weeks later, as per PCWG3, or death from any cause in the absence of progression. Participants who do not progress or die including those who withdraw from the study or are lost to follow-up will be censored at the time of last valid PSA measurement.
Time Frame: From the randomization up to 23 months
Population: All participants from the ITT analysis set. Number of participants censored in [Lu-177]-PNT2002 (Arm A)=133, Abiraterone or Enzalutamide (Arm B)=54. The "Overall Number of Participants Analyzed" reported is inclusive of the censored participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomization Phase: [Lu-177]-PNT2002 (Arm A) | Randomization Phase: Abiraterone or Enzalutamide (Arm B)
Number analyzed (Participants) | 276 | 136
months | 7.0 [4.8 to 9.9] | 3.9 [3.5 to 4.3]

6. Secondary Outcome: Overall Survival
Description: Time from the date of randomization until death due to any cause.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2029-03

ADVERSE EVENTS:
Time Frame: Baseline up to 26 months
Description: All participants from the safety analysis set were included in reporting of serious and other (not including serious) adverse events. For all-cause mortality reporting, all participants in the study were included.
Groups:
- Dosimetry Phase: [Lu-177]-PNT2002: Participants received 6.8 GBq (±10%) of [Lu-177]-PNT2002 every 8 weeks for 4 cycles.
- Randomization Phase: Abiraterone or Enzalutamide (Arm B) / Abiraterone or Enzalutamide: Participants received either of below treatments until radiographic progression.
  * Enzalutamide 160 mg orally once daily (or)
  * Abiraterone 1000 mg orally once daily coadministered with prednisone 5 mg orally twice daily or dexamethasone 0.5 mg orally once daily.
- Randomization Phase: Abiraterone or Enzalutamide (Arm B) / [Lu-177]-PNT2002: Arm B participants who experienced radiographic progression per BICR (or after final OS, per local investigator-assessment), had not started an intervening treatment, and had no uncontrolled AEs were eligible to consent to cross over to receive 6.8 GBq (±10%) of [Lu-177]-PNT2002 intravenous infusion every 8 weeks for 4 cycles.
Arm/Group | Dosimetry Phase: [Lu-177]-PNT2002 | Randomization Phase: [Lu-177]-PNT2002 (Arm A) | Randomization Phase: Abiraterone or Enzalutamide (Arm B) / Abiraterone or Enzalutamide | Randomization Phase: Abiraterone or Enzalutamide (Arm B) / [Lu-177]-PNT2002 | PK Extension Phase: [Lu-177]-PNT2002
All-Cause Mortality (participants affected / at risk) | 13/27 | 76/276 | 32/136 | 12/77 | 0/16
Serious Adverse Events (participants affected / at risk) | 6/27 | 47/269 | 30/130 | 14/77 | 2/15
Other Adverse Events (participants affected / at risk) | 24/27 | 259/269 | 117/130 | 59/77 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dosimetry Phase: [Lu-177]-PNT2002 (N=27) | Randomization Phase: [Lu-177]-PNT2002 (Arm A) (N=269) | Randomization Phase: Abiraterone or Enzalutamide (Arm B) / Abiraterone or Enzalutamide (N=130) | Randomization Phase: Abiraterone or Enzalutamide (Arm B) / [Lu-177]-PNT2002 (N=77) | PK Extension Phase: [Lu-177]-PNT2002 (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 2 (3) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathy alcoholic (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 1 (2) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ecg signs of myocardial ischaemia (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urothelium erosion (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gangrene (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dosimetry Phase: [Lu-177]-PNT2002 (N=27) | Randomization Phase: [Lu-177]-PNT2002 (Arm A) (N=269) | Randomization Phase: Abiraterone or Enzalutamide (Arm B) / Abiraterone or Enzalutamide (N=130) | Randomization Phase: Abiraterone or Enzalutamide (Arm B) / [Lu-177]-PNT2002 (N=77) | PK Extension Phase: [Lu-177]-PNT2002 (N=15)
Anaemia (Blood and lymphatic system disorders) | 6 (16) | 48 (78) | 13 (25) | 14 (25) | 4 (4)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 5 (9) | 3 (5) | 1 (1) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 9 (12) | 1 (2) | 2 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (4) | 5 (5) | 1 (1) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3) | 8 (14) | 1 (1) | 2 (4) | 3 (5)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 11 (14) | 6 (7) | 3 (3) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (4) | 54 (62) | 23 (25) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 40 (46) | 13 (18) | 6 (6) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 7 (7) | 100 (116) | 2 (2) | 19 (23) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 5 (5) | 2 (2) | 2 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (8) | 84 (105) | 25 (28) | 17 (23) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 28 (33) | 6 (6) | 6 (9) | 0 (0)
Asthenia (General disorders) | 1 (1) | 14 (17) | 6 (11) | 2 (3) | 0 (0)
Chest pain (General disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Fatigue (General disorders) | 8 (10) | 144 (184) | 52 (62) | 24 (30) | 7 (8)
Feeling abnormal (General disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 15 (18) | 4 (4) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 30 (33) | 8 (8) | 5 (5) | 3 (3)
Pain (General disorders) | 0 (0) | 7 (7) | 6 (6) | 3 (5) | 1 (1)
Covid-19 (Infections and infestations) | 2 (2) | 27 (28) | 10 (11) | 2 (2) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 12 (21) | 7 (9) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 20 (21) | 9 (13) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (5) | 1 (1) | 1 (1) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 6 (9) | 2 (4) | 1 (2) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 15 (19) | 5 (5) | 5 (5) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2) | 18 (23) | 4 (4) | 2 (2) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 8 (20) | 1 (1) | 0 (0) | 4 (8)
Sputum abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 17 (21) | 16 (21) | 7 (10) | 2 (2)
Weight increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
White blood cell count decreased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 40 (46) | 17 (17) | 8 (10) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 9 (9) | 4 (4) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (8) | 0 (0) | 3 (3) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (6) | 7 (7) | 2 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 2 (2) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (6) | 7 (9) | 3 (3) | 3 (4) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 6 (9) | 5 (7) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 75 (95) | 35 (48) | 15 (18) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 56 (66) | 28 (36) | 8 (12) | 2 (2)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 13 (15) | 6 (8) | 3 (4) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 16 (19) | 10 (10) | 3 (3) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (7) | 3 (4) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 29 (32) | 17 (20) | 6 (6) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 18 (21) | 11 (12) | 6 (8) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2) | 6 (6) | 0 (0) | 5 (5) | 2 (2)
Headache (Nervous system disorders) | 3 (4) | 20 (25) | 10 (10) | 3 (3) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 6 (6) | 4 (5) | 1 (1) | 2 (2)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 4 (4) | 3 (3) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 6 (6) | 5 (6) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (2) | 12 (12) | 13 (15) | 4 (4) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 6 (8) | 1 (1) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 3 (3) | 12 (13) | 6 (12) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 1 (2)
Urothelium erosion (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 24 (25) | 6 (6) | 5 (5) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 16 (19) | 5 (6) | 5 (5) | 2 (2)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 11 (12) | 17 (18) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 8 (15) | 13 (20) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2025-07-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT04647526/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-26): https://cdn.clinicaltrials.gov/large-docs/26/NCT04647526/SAP_001.pdf